CLINICAL TRIAL: NCT03544827
Title: The Effects of Low Dose Atropine on Choroidal Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Franklin Bui, Co-principal investigator, State University of New York College of Optometry
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1168531-2
Record Dates: First submitted 2018-05-08; First posted 2018-06-04 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Myopia
Keywords: Atropine
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and main investigator will be blinded to the allocation concealment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atropine 0.01% then atropine 0.1% (Experimental): Participants will be on topical atropine 0.01% ophthalmic solution QD OU for 1 week (7 days) and then topical atropine 0.1% ophthalmic solution QD OU for 1 week (7 days) with a washout period of 4 weeks in between each intervention
  Interventions: Drug: Atropine
- Atropine 0.1% then atropine 0.01% (Experimental): Participants will be on topical atropine 0.1% ophthalmic solution QD OU for 1 week (7 days) and then topical atropine 0.01% ophthalmic solution QD OU for 1 week (7 days) with a washout period of 4 weeks in between each intervention
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Atropine 0.01% then atropine 0.1%
  Other Names: Atropine 0.01%; Atropine 0.1%
Drug: Atropine — Atropine 0.1% then atropine 0.01%
  Other Names: Atropine 0.1%; Atropine 0.01%

SUMMARY:
Atropine eye drops are considered to be an effective form of myopia control in human eyes. However, the mechanism by which it exerts it effects are not fully understood. Thickening of the choroid subsequent to atropine administration may play an important role in the mechanisms by which atropine induces myopia control. Literature also notes that choroidal thickness undergoes diurnal variations, which is a variable that will be controlled in this study in order to examine atropine's effects on different baseline choroidal thicknesses.

The purpose of the proposed study is to characterize better the influence of atropine on choroid thickness. The study aims are to:

1. Determine the effect of low dose concentration of topical atropine (0.1% and 0.01%) on choroid thickness
2. Determine the effect of topical atropine on choroid thickness in relationship to baseline thickness throughout the day and after one week of daily instillation

Hypothesis: Atropine's effect on choroidal thickness will be dependent on the subject's baseline thickness measurements, at a designated time of the day when the choroid is at its thinnest.

DETAILED DESCRIPTION:
Atropine eye drops are an effective form of myopia control in children with progressive myopia1, but the mechanism in which this occurs is still not fully understood.

The choroid has been established to play a significant role in the modulation of ocular growth in the chick eye;2 eyes with thicker choroids grow slower than eyes with thinner choroids.3 Choroidal compensation has also been discovered in other animal species including tree shrews,4 marmosets,5 rhesus macaques,6 guinea pigs,7, 8 and even in humans.9, 10 A study in humans demonstrated how the thickening of the choroid subsequent to atropine use may contribute to the mechanisms by which atropine induces myopia control.11 These results are supported by another study where children with less choroidal thickening over time exhibited faster axial growth.12 Furthermore, diurnal variation in choroidal thickness has been documented13, 14 and individuals with thinner choroids exhibited less variation in thickness across the day. 13

Currently, atropine is prescribed by eye care providers on a daily basis and administered at night for convenience. However, choroidal thickness undergoes diurnal variations13, and the efficacy of atropine on myopia control in relationship to the patient's baseline choroidal thickness is unknown.

A preliminary study shows that atropine 1% has an effect on reducing choroidal thinning throughout the day, but how this translates to low concentration atropine as is commonly prescribed in myopia control treatment is unknown. Specifically, preliminary results reveal that the maximal pharmaceutical effects on choroidal thickening occurred one hour after atropine 1% instillation in the morning, but its relative efficacy during specific time points and duration of the day is still unclear. Also, baseline diurnal measurements demonstrate that the choroid thins in the morning, is thinnest at noon, and gradually thickens in the evening and overnight. The effects of atropine on the choroid from noon to the afternoon were not explicitly measured in our previous study, and therefore, are measurements of interest. While it is critical to understand the effects of low dose atropine on choroidal thickness throughout the evening as commonly prescribed clinically, it is important to also understand its effects when the choroid is shown to thin during the day. Additionally, the study measured changes in choroidal thickness after one instillation of atropine, but did not explore the effects of daily instillation on choroidal thickness and whether there is further minimization of choroidal thinning.

Thus, the objective of this study is to provide data to characterize the influence of low dose atropine on choroid thickness. The study aims are:

1. To determine the effect of low dose topical atropine (0.1% and 0.01%) on choroid thickness
2. To determine the effect of topical atropine on choroid thickness in relationship to baseline thickness throughout the day and after one week of daily instillation.

It is hypothesized that atropine's effect on choroidal thickness will be dependent on the subject's baseline thickness measurements, at a designated time of the day when the choroid is at its thinnest.

Potential risks of this study are related to the use of atropine eye drops. Atropine 0.1% and 0.01% eye drops may cause dilation of the pupil (mydriasis) and paralysis of accommodation (cycloplegia).15 There are also rare ocular and systemic adverse effects associated with the use of atropine eye drops as described in section C3 below.15 However, using the minimum dosage in combination with low concentrations of the drug will minimize these adverse effects associated with atropine.16 Participants will be asked if they have experienced any reactions to eye drops in the past. The puncta can be occluded as a preventative measure against systemic absorption. Risks can be further minimized by preparing for adverse systemic side effects and by immediate recognition of the signs and appropriate monitoring. The participant will also be educated to report any unforeseen side effects from instillation of the atropine according to the instructions detailed in consent form. All participants will be trained to promptly report any side effects to the investigators.

Medline and Pubmed databases were used for literature review.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 - 35 years
* Good general and ocular health
* Soft contact lens wearers to cease lens wear for at least 24 hours
* No previous rigid gas permeable lens wear
* Not taking monoamine oxidase inhibitors (MAOIs) and are not pregnant

Exclusion Criteria:

* History of ocular surgery, including refractive surgery
* Use of ocular medications
* Amblyopia
* Conditions where topical atropine is contraindicated
* Any eye or systemic disease that affect vision or refractive error

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  Measure choroidal thickness changes at baseline and compare to choroidal thickness after intervention of atropine 0.01% and atropine 0.1%

SECONDARY OUTCOMES:
Visual acuity | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  Measure distance and near visual acuity at baseline and re-measure after intervention of atropine 0.01% and atropine 0.1% for any changes
Axial length | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  Measure axial length at baseline and compare to changes after intervention of atropine 0.01% and atropine 0.1%
Lens thickness | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  Measure lens thickness at baseline and compare to changes after intervention of atropine 0.01% and atropine 0.1%
Anterior chamber depth | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  Measure anterior chamber depth at baseline and compare to changes after intervention of atropine 0.01% and atropine 0.1%
Quality of Vision (QoV) Questionnaire | 1 hour, 4 hours, 8 hours, and 1 week from baseline measurement
  The questionnaire is a Rasch-tested, linear-scaled, 30-item instrument on three scales providing a QoV score in terms of symptom frequency, severity, and bothersome. There are four options of increasing severity of symptoms from none, mild, moderate, and to severe for each item. The use of Rasch analysis turns the original questionnaire responses (raw ordinal data) into continuous interval data, providing a linear measurement; it is on a linear interval scale.
Tear break up time (TBUT) | Baseline and 1 week from baseline measurement
  Sodium fluorescein dye is added to the eye and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop; compare any differences between baseline and after one week of atropine use
Schirmer strip test | Baseline and 1 week from baseline measurement
  Measure amount of tear production; compare value at baseline to values after 1 week of atropine use to determine if tear production is affected with atropine use
Ocular Surface Disease Index (OSDI) | Baseline and 1 week from baseline measurement
  This is a 12-item questionnaire with 5 options from 0 to 5 (with 0 indicating none of the time, and increases to 5 indicating all of the time). The sum of the scores across the 12 items are totaled, and inputted into a formula to generate a sliding scale of the disease condition. The scale ranges from 0 to 100, with higher scores representing greater disability of the disease condition. This questionnaire will be completed at baseline and after 1 week of atropine use to compare for any differences.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Benavente-Perez, PhD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY College of Optometry, New York, New York, United States

REFERENCES:
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Wallman J, Winawer J. Homeostasis of eye growth and the question of myopia. Neuron. 2004 Aug 19;43(4):447-68. doi: 10.1016/j.neuron.2004.08.008. PMID 15312645
- [Background] Nickla DL, Totonelly K. Choroidal thickness predicts ocular growth in normal chicks but not in eyes with experimentally altered growth. Clin Exp Optom. 2015 Nov;98(6):564-70. doi: 10.1111/cxo.12317. PMID 26769180
- [Background] Siegwart JT Jr, Norton TT. The susceptible period for deprivation-induced myopia in tree shrew. Vision Res. 1998 Nov;38(22):3505-15. doi: 10.1016/s0042-6989(98)00053-4. PMID 9893785
- [Background] Troilo D, Nickla DL, Wildsoet CF. Choroidal thickness changes during altered eye growth and refractive state in a primate. Invest Ophthalmol Vis Sci. 2000 May;41(6):1249-58. PMID 10798638
- [Background] Hung LF, Wallman J, Smith EL 3rd. Vision-dependent changes in the choroidal thickness of macaque monkeys. Invest Ophthalmol Vis Sci. 2000 May;41(6):1259-69. PMID 10798639
- [Background] Howlett MH, McFadden SA. Form-deprivation myopia in the guinea pig (Cavia porcellus). Vision Res. 2006 Jan;46(1-2):267-83. doi: 10.1016/j.visres.2005.06.036. Epub 2005 Aug 31. PMID 16139323
- [Background] Howlett MH, McFadden SA. Spectacle lens compensation in the pigmented guinea pig. Vision Res. 2009 Jan;49(2):219-27. doi: 10.1016/j.visres.2008.10.008. Epub 2008 Dec 4. PMID 18992765
- [Background] Woodman EC, Read SA, Collins MJ. Axial length and choroidal thickness changes accompanying prolonged accommodation in myopes and emmetropes. Vision Res. 2012 Nov 1;72:34-41. doi: 10.1016/j.visres.2012.09.009. Epub 2012 Sep 24. PMID 23017772
- [Background] Chakraborty R, Read SA, Collins MJ. Monocular myopic defocus and daily changes in axial length and choroidal thickness of human eyes. Exp Eye Res. 2012 Oct;103:47-54. doi: 10.1016/j.exer.2012.08.002. Epub 2012 Aug 16. PMID 22971342
- [Background] Zhang Z, Zhou Y, Xie Z, Chen T, Gu Y, Lu S, Wu Z. The effect of topical atropine on the choroidal thickness of healthy children. Sci Rep. 2016 Oct 7;6:34936. doi: 10.1038/srep34936. PMID 27713535
- [Background] Read SA, Alonso-Caneiro D, Vincent SJ, Collins MJ. Longitudinal changes in choroidal thickness and eye growth in childhood. Invest Ophthalmol Vis Sci. 2015 May;56(5):3103-12. doi: 10.1167/iovs.15-16446. PMID 26024094
- [Background] Tan CS, Ouyang Y, Ruiz H, Sadda SR. Diurnal variation of choroidal thickness in normal, healthy subjects measured by spectral domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Jan 25;53(1):261-6. doi: 10.1167/iovs.11-8782. PMID 22167095
- [Background] Chakraborty R, Read SA, Collins MJ. Diurnal variations in axial length, choroidal thickness, intraocular pressure, and ocular biometrics. Invest Ophthalmol Vis Sci. 2011 Jul 11;52(8):5121-9. doi: 10.1167/iovs.11-7364. PMID 21571673
- [Background] North RV, Kelly ME. A review of the uses and adverse effects of topical administration of atropine. Ophthalmic Physiol Opt. 1987;7(2):109-14. doi: 10.1111/j.1475-1313.1987.tb01004.x. PMID 2958765
- [Background] Gong Q, Janowski M, Luo M, Wei H, Chen B, Yang G, Liu L. Efficacy and Adverse Effects of Atropine in Childhood Myopia: A Meta-analysis. JAMA Ophthalmol. 2017 Jun 1;135(6):624-630. doi: 10.1001/jamaophthalmol.2017.1091. PMID 28494063
- [Background] Pediatric Eye Disease Investigator Group.. A randomized trial of atropine vs. patching for treatment of moderate amblyopia in children. Arch Ophthalmol. 2002 Mar;120(3):268-78. doi: 10.1001/archopht.120.3.268. PMID 11879129
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] Rahman W, Chen FK, Yeoh J, Patel P, Tufail A, Da Cruz L. Repeatability of manual subfoveal choroidal thickness measurements in healthy subjects using the technique of enhanced depth imaging optical coherence tomography. Invest Ophthalmol Vis Sci. 2011 Apr 8;52(5):2267-71. doi: 10.1167/iovs.10-6024. Print 2011 Apr. PMID 21087970